CLINICAL TRIAL: NCT04858438
Title: Pain After Insufflation for Robotic Sacrocolpopexy (PAIRS) Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1716019
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Sacrocolpopexy; Pneumoperitoneum; Postoperative pain
MeSH Terms: conditions — Pelvic Organ Prolapse; Pneumoperitoneum; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either standard pneumoperitoneum (15 mmHg) versus a lower level of pneumoperitoneum (12 mmHg).
Who Masked: Participant
Masking Description: Patients will be unaware of their study group status and unaware of level of pneumoperitoneum used during their surgical procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Insufflation Group (Active Comparator): Patients will receive standard insufflation during surgery (15 mm Hg).
  Interventions: Procedure: Insufflation during surgery
- Low Insufflation Group (Experimental): Patients will receive a lower level of insufflation during surgery (12 mm Hg or lower).
  Interventions: Procedure: Insufflation during surgery

INTERVENTIONS:
Procedure: Insufflation during surgery — This is the amount of insufflation using during the surgical procedure.

SUMMARY:
This study evaluates post-operative pain between different insufflation pressures during robotic-assisted sacrocolpopexy. Subjective pain and narcotic usage after surgery will be measured.

DETAILED DESCRIPTION:
This is a prospective single-blind randomized controlled trial of adult women undergoing robotic-assisted sacrocolpopexy for pelvic organ prolapse. Each surgery will be performed by a board-certified Female Pelvic Medicine & Reconstructive Surgery (FPMRS) surgeon with a standard technique other than pneumoperitoneum level. A sacrocolpopexy for apical prolapse may be performed at the same time as a hysterectomy and other clinically indicated procedures if desired by the patient and as part of the standard of care. Patients will be stratified by hysterectomy prior to randomization. Postoperatively, patients will be evaluated with a Visual Analogue Scale (VAS) as well as prescribed narcotic analgesic use and followed up to 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to have a robotic-assisted sacrocolpopexy surgery for pelvic organ prolapse.
* Age 18-90 years
* Can read and understand the consent form and consents to the procedure

Exclusion Criteria:

* Patients undergoing other procedures
* Patients who do not consent to participate.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This procedure only applies to women.
Enrollment: 80 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pain on a visual analogue scale, ranging from 1-10 with a higher score meaning more pain. | Pain will be assessed within 24 hours of the surgery. .
  Pain will be assessed during the 24-hour post-operative period.
Post-operative Pain on a visual analogue scale, ranging from 1-10 with a higher score meaning more pain. | Pain will be assessed at the two-week post-operative follow-up visit.
  Pain will be assessed during the two-week post-operative period.
Safety using Operation length, blood loss, need to increase insufflation, operative conversion rates. These are all counts with higher numbers meaning worse outcomes. | Safety will be assessed during the procedure.
  The safety of the lower insufflation pressure will be assessed during the procedure.
Safety using Operation length, blood loss, need to increase insufflation, operative conversion rates. These are all counts with higher numbers meaning worse outcomes. | Safety will be assessed immediately post-operatively.
  The safety of the lower insufflation pressure will be assessed immediately post-operatively.
Safety using Operation length, blood loss, need to increase insufflation, operative conversion rates. These are all counts with higher numbers meaning worse outcomes. | Safety will be assessed at the two-week follow-up visit.
  The safety of the lower insufflation pressure will be assessed at the two-week follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension St. John Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rustia GM, Baracy MG Jr, Khair E, Hagglund KH, Aslam MF. Pain With Differing Insufflation Pressures During Robotic Sacrocolpopexy: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jul 1;142(1):151-159. doi: 10.1097/AOG.0000000000005231. Epub 2023 Jun 7. PMID 37348093